CLINICAL TRIAL: NCT06373289
Title: Target Oxygen Saturation Ranges in Infants With Bronchopulmonary Dysplasia Associated Pulmonary Hypertension
Brief Title: Pulmonary Hypertension and Oxygen Saturation Targeting in Preterm Infants
Acronym: PHOX
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Samuel Gentle, Assistant Professor, Yale University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 000539476; 1K23HD113837-01A1 (NIH)
Record Dates: First submitted 2024-03-19; First posted 2024-04-18 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Bronchopulmonary Dysplasia; Pulmonary Hypertension
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Hypertension, Pulmonary

STUDY DESIGN:
Intervention Model Description: Single center, randomized cross-over pilot study with a 1:1 parallel allocation of infants to SpO2 targets of 92-95% (control) and 95-98% (intervention) using a stratified permuted block design. Following 1 week of exposure A, infants will cross over to exposure B for 1 week with a 1-week washout period.
Who Masked: Outcomes Assessor
Masking Description: The PI will perform bedside echocardiography precluding masking to group allocation. All echocardiograms will be further reviewed by a cardiologist masked to group allocation with additional cardiologist review in instances of disagreement. Inter-rater reliability testing will also be performed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oxygen saturation target 92-95% (Active Comparator): At UAB and Yale oxygen saturation targeting is achieved using systematic oxygen saturation histogram monitoring every 3-4 hours by nurse, respiratory therapists, and physicians. Upon randomization to this arm, infants oxygen saturation alarm limits will be adjusted to 92-95% after which an FiO2 modification algorithm will be employed to maintain targets. Daily compliance reports will be generated to ensure oxygen saturation achievement corresponds with oxygen saturation targets. Infants will be exposed to a 1 week period after which they will crossover to the alternative oxygen saturation target with a 1 week washout period in between targets.
  Interventions: Device: lower oxygen saturation target using Nellcor pulse oximetry sensors
- Oxygen saturation target 95-98% (Active Comparator): At UAB and Yale oxygen saturation targeting is achieved using systematic oxygen saturation histogram monitoring every 3-4 hours by nurse, respiratory therapists, and physicians. Upon randomization to this arm, infants oxygen saturation alarm limits will be adjusted to 95-98% after which an FiO2 modification algorithm will be employed to maintain targets. Daily compliance reports will be generated to ensure oxygen saturation achievement corresponds with oxygen saturation targets. Infants will be exposed for a 1 week period after which they will crossover to the alternative oxygen saturation target with a 1 week washout period in between targets.
  Interventions: Device: higher oxygen saturation target using Nellcor pulse oximetry sensors

INTERVENTIONS:
Device: higher oxygen saturation target using Nellcor pulse oximetry sensors — The intervention will be a cross over exposure to the higher oxygen saturation target.
  Arms: Oxygen saturation target 95-98%
Device: lower oxygen saturation target using Nellcor pulse oximetry sensors — The intervention will be a cross over exposure to the lower oxygen saturation target.
  Arms: Oxygen saturation target 92-95%

SUMMARY:
Around 50% of infants born extremely preterm develop a chronic lung disease known as bronchopulmonary dysplasia of which some infants will also develop pulmonary hypertension of which 50% of children will die before the age of 2. Physicians are currently limited in their ability to select the most appropriate oxygen targets that will improve outcomes in infants with this condition. This clinical trial will determine whether using different amounts of oxygen improve outcomes in infants with this disease.

DETAILED DESCRIPTION:
Infants born between 22.0 to 31.6 weeks' gestational age with bronchopulmonary dysplasia associated pulmonary hypertension, are receiving supplemental oxygen, and have mature retinas will be randomized to SpO2 targets of either (1) 92-95% (control) or (2) 95-98% (intervention).

Using a cross over design with a 1:1 parallel allocation of infants randomized using a stratified permuted block design. Following 1week of exposure A, infants will cross over to exposure B for 1 week with a 1-week washout period. Bedside providers will follow pre-specified algorithms to maintain oxygen targets during the randomization period. Reports of oxygen saturation performance will also be provided to bedside providers through oxygen saturation histograms.

ELIGIBILITY:
Inclusion Criteria:

* Between 22w 0/7d and 31w 6/7d gestation at birth
* Diagnosed with echocardiographic pulmonary hypertension (1) >20% flow of blood across the PDA from the pulmonary to arterial circulation, (2) end-systolic flattening of the interventricular septum (eccentricity index >1.3), or (3) right ventricular pressure estimates ≥ 35 mm Hg
* Receiving supplemental oxygen
* Have mature retinas

Exclusion Criteria:

* Major congenital anomalies

Ages: 1 Month to 5 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 39 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2029-07-01 (Estimated); Study Completion 2030-07-01 (Estimated)

PRIMARY OUTCOMES:
Intermittent hypoxemia event duration | From date of randomization until 3 weeks have elapsed or date of discharge, whichever came first
  The average duration of time (in seconds) an infant's oxygen saturation decrease below 80%.

SECONDARY OUTCOMES:
Echocardiographic shunting | through study completion, 3 weeks from date of randomization until 3 weeks have elapsed or date of discharge, whichever came first
  >20% flow of blood across the PDA from the pulmonary to arterial circulation
Echocardiographic interventricular septal flattening | From date of randomization until 3 weeks have elapsed or date of discharge, whichever came first
  End-systolic flattening of the interventricular septum (eccentricity index >1.3)
Echocardiographic tricuspid regurgitation | From date of randomization until 3 weeks have elapsed or date of discharge, whichever came first
  Right ventricular pressure estimates
Intermittent hypoxemia frequency | From date of randomization until 3 weeks have elapsed or date of discharge, whichever came first
  Number of daily events during which an infant's oxygen saturation decreases below 80%
Cumulative hypoxemia | From date of randomization until 3 weeks have elapsed or date of discharge, whichever came first
  Daily duration during which an infant's oxygen saturation is <80%
Brain natriuretic peptide | From date of randomization until 3 weeks have elapsed or date of discharge, whichever came first
  A polypeptide released from the cardiac ventricles indicative of right heart strain

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Gentle, Principal Investigator — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Yale New Haven Hospital, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No